CLINICAL TRIAL: NCT07226869
Title: Computer Guided Microwave Liver Ablation
Acronym: MWA Sim
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NE Scientific INC (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Dartmouth-Hitchcock Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NES_2025_01; 1R44CA287803-01 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; liver neoplasm; primary liver cancer; microwave ablation (MWA); percutaneous ablation; computer-assisted ablation; simulation-guided ablation; 3D ablation planning; treatment planning software; image-guided ablation; local tumor progression
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Masking Description: Imaging outcomes will be assessed by independent radiologists blinded to intervention status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Computerized Guidance (Experimental): Patients enrolled in this arm will undergo liver cancer microwave ablation under computerized guidance.
  Interventions: Device: Computer-Assisted Microwave Liver Ablation

INTERVENTIONS:
Device: Computer-Assisted Microwave Liver Ablation — Computer-assisted image-processing software used intraoperatively to assist in percutaneous thermal ablation. The software performs segmentation and registration of pre-procedural and intraprocedural imaging, and simulates the expected ablation zone based on probe position, applied energy, and adjacent vascular structures. The output is displayed in 3D multiplanar images to be used by the treating physician to assist in planning, targeting, and intraprocedural decision-making regarding adequacy of ablation coverage. After each ablation activation, the treating physician determines registration accuracy and decides whether any additional ablation is required, based on images of the software estimation of what tissues have and have not been treated.

SUMMARY:
The goal of this clinical trial is to learn if the intraoperative use of a computer guidance software can improve the success of liver tumor ablation in adults. The employed software calculates and displays a simulation of the ablation such that the physician can visualize what portion of the target tumor has, and has not been treated at any point during the procedure. The main questions it aims to answer are: 1) Does the use of the computer guidance software reduce the number of times a tumor is incompletely treated. 2) Does the use of the computer guidance software reduce the rate of local tumor recurrence at 2 year follow-up? 3) Was there an increase or a decrease in medical problems for participants after a procedure where the guidance software was used?

Researchers will compare liver tumor treatment using the computer guidance software with an historic control to see if the addition of the guidance software improved the outcomes after an ablation.

Participants will:

Undergo CT-guided microwave ablation treatment of a liver tumor using computer-assisted simulation. Visit the clinic at one month and then every 3 months for blood tests and a contrast-enhanced CT or MRI imaging study (as per standard of care)

DETAILED DESCRIPTION:
Accublate (NE Scientific, Inc) is a computer-based tumor ablation guidance software that uniquely provides real-time simulation of expected ablation volumes. In a previously reported study of Radiofrequency Ablation, the improved visualization of treated versus untreated target tumor was associated with improved outcomes. This study examines clinical application of the simulation software for microwave ablation (MWA), which will be evaluated in a 24 month two-center clinical trial.

At Dartmouth Hitchcock Medical Center (DHMC), and at one other hospital, under IRB approval, adults referred from local Liver Tumor Boards for curative local treatment of up to four Hepatocellular Carcinoma (HCC) tumors of 2-5 cm diameter will be offered participation.

After providing informed consent, and meeting inclusion and exclusion criteria, the CT-guided MWA ablation will be performed, with the physician having the benefit of the graphical display of the Accublate MWA simulation guidance software. Prior to the ablation, the software provides 3D graphical display for planning, that includes the tumor, desired margin, and interactive model of the ablation probe and superimposed expected ablation volume at particular energy settings. During placement, the software permits registration of updated image of the actual probe position to original image of the segmented tumor, and with the interactive ablation volume settings, allows assessment of adequacy of targeting. After each activation of the ablation, the calculated simulated ablation volume is provided to indicate what tissues have, and have not, been ablated. These 3D views then provide guidance for intraprocedural adjustments to ensure target coverage by overlapping ablations, if indicated.

Patients are routinely admitted for overnight observation and receive IV pain and nausea medication if needed. One month after the ablation, patients will have a follow-up outpatient contrast-enhanced abdominal CT, and from these images, the rate of complete ablation (Technical Efficacy) will be determined. Additionally, patients will be followed at 3 month intervals for 24 months after the ablation to detect any complications, tumor recurrence (Local Tumor Progression), and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, with life expectancy of at least 1 year
2. Diagnosis of hepatocellular carcinoma (HCC) confirmed by:

   * LI-RADS 5 imaging features or
   * Histopathology
   * Cirrhosis with AFP > 400
3. Localized disease without macrovascular invasion or extrahepatic metastasis, eligible for curative-intent percutaneous thermal ablation, defined as:

   o Up to 5 lesions with at least one lesion, 2 -5 cm, and no lesion >5 cm diameter
4. Tumor location deemed technically feasible for percutaneous ablation by the treating interventional radiologist
5. ECOG Performance Status 0-2
6. Adequate coagulation status, defined as:

   * Platelets ≥ 50,000/μL
   * INR ≤ 1.8 (or correctable)
7. Ability to undergo contrast-enhanced CT or MRI
8. Willingness and ability to provide informed consent

Exclusion Criteria:

1. Prior local therapy to the target lesion (ablation, TACE, SBRT, or resection) or to a lesion within 1 cm of the target lesion
2. More than 5 hepatic lesions, or any lesion ineligible for technically complete ablation
3. uncontrolled hepatic decompensation, including:

   o Persistent encephalopathy
4. Uncorrectable coagulopathy or contraindication to percutaneous liver intervention
5. Contraindication to contrast-enhanced imaging (e.g., severe CKD without dialysis, contrast allergy not correctable with premedication)
6. Active systemic infection
7. Pregnancy
8. Inability to comply with follow-up imaging schedule

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2030-03-02 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Local Tumor Progression | Assessed at each imaging follow-up visit ( at every 3 months, up to 24 months).
  Local Tumor Progression (LTP) is defined as the appearance of new or enlarging nodular or irregular arterial phase enhancement with washout at or within the edge of a previously ablated lesion after an earlier imaging study has demonstrated complete ablation (technical effectiveness). LTP is determined on serial contrast-enhanced CT or MRI according to LI-RADS treatment response criteria or equivalent institutional standards.
Technical Effectiveness | 1 month post-procedure
  Technical Effectiveness is defined as complete ablation of all target tumor tissue, demonstrated by the absence of any nodular or irregular arterial phase enhancement within or along the margin of the ablation zone on the first post-ablation contrast-enhanced imaging study (CT or MRI). This assessment is performed approximately one month after the procedure. Imaging is interpreted according to LI-RADS treatment response criteria (LR-TR) or equivalent institutional criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Borsic, PHD, Study Director — NE Scientific INC
Locations (1):
- Dartmouth HItchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the published results, including key clinical, imaging, and procedural variables relevant to study outcomes.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 12 months after publication of the primary study results and continuing for a minimum of 5 years thereafter.
Access Criteria: Qualified investigators affiliated with academic, research, or healthcare institutions. For research purposes consistent with the scientific aims of the original study or for meta-analyses addressing related clinical or technical questions. Study protocol, statistical analysis plan, and data dictionary will be available upon reasonable request. Requests for de-identified data may be submitted to the Principal Investigator (Dr. Eric Hoffer, Dartmouth-Hitchcock Medical Center) by email. Access will be granted following review of the request and execution of a data use agreement approved by the sponsor (NE Scientific, Inc.) and the Principal Investigator.

REFERENCES:
- [Background] Hoffer EK, Borsic A, Patel SD. Validation of Software for Patient-Specific Real-Time Simulation of Hepatic Radiofrequency Ablation. Acad Radiol. 2022 Oct;29(10):e219-e227. doi: 10.1016/j.acra.2021.12.018. Epub 2022 Jan 14. PMID 35039220
- [Background] Hoffer EK, Drinane MC, Bhatnagar V, Mehta R, Munger DP, Borsic A. Radiofrequency ablation of hepatocellular carcinoma guided by real-time physics-based ablation simulation: a prospective study. Int J Hyperthermia. 2024;41(1):2331704. doi: 10.1080/02656736.2024.2331704. Epub 2024 Mar 19. PMID 38503326